CLINICAL TRIAL: NCT07136922
Title: First in Human Safety and Ease of Use Assessment of 400mg Progesterone Callavid in Women With Luteal Phase Insufficiency
Acronym: FREEDOM
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Calla Lily Clinical Care Ltd (Industry)
Collaborators: University Hospitals Coventry and Warwickshire NHS Trust (Other); University of Warwick (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SQ641924
Record Dates: First submitted 2025-07-28; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Luteal Phase Insuffiency; Progesterone Delivery
Keywords: progesterone delivery; progesterone; vaginal drug delivery; callavid; cyclogest; women's health
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Intervention Model Description: The trial consists of three rounds, conducted over three consecutive menstrual cycles. Participants are randomised to receive either Cyclogest 400mg progesterone pessary in the first round, crossing over to 400mg progesterone Callavid (administered for 2 hours) in the second round, or 400mg progesterone Callavid (administered for 2 hours) in the first round crossing over to Cyclogest 400mg progesterone pessary in the second round.
  The third round is to investigate the safety of 400mg progesterone Callavid when administered for 3 hours. This would inform us on the safety of the additional hour of wear time. Each arm will complete the third round following the first two crossover rounds.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Callavid 2-hr first, Cyclogest second, Callavid 3-hr third (Active Comparator): Participants are randomised to use Callavid first for 2 hour wear before crossing over to use Cyclogest. In the third round, participants receive Callavid again but for 3 hour wear.
  Interventions: Combination Product: 400mg progesterone Callavid - 2hr wear; Drug: Cyclogest 400 mg; Combination Product: 400mg progesterone Callavid - 3hr wear
- Cyclogest first, Callavid 2-hr second, Callavid 3-hr third (Active Comparator): Participants are randomised to use Cyclogest first before crossing over to use Callavid for 2 hour wear. In the third round, participants receive Callavid again but for 3 hour wear.
  Interventions: Combination Product: 400mg progesterone Callavid - 2hr wear; Drug: Cyclogest 400 mg; Combination Product: 400mg progesterone Callavid - 3hr wear

INTERVENTIONS:
Combination Product: 400mg progesterone Callavid - 2hr wear — 400mg progesterone Callavid, 2 hour wear, twice daily for 7 days
Drug: Cyclogest 400 mg — Cyclogest 400 mg pessary, twice daily for 7 days
Combination Product: 400mg progesterone Callavid - 3hr wear — 400mg progesterone Callavid, 3 hour wear, twice daily for 7 days

SUMMARY:
The aim of this clinical trial is to assess safety of a new vaginal 400mg progesterone drug-device combination product in a first in human trial. Additionally, it aims to assess user acceptability and ability to deliver progesterone. This Phase I trial is a randomised open-label first-in-human crossover trial, recruiting participants who are non-pregnant with luteal phase insufficiency. The main questions it aims to answer are:

1. What are the safety and tolerability profiles of the two progesterone formulations (400mg Progesterone Callavid vs. Cyclogest 400 mg), including the incidence of adverse events (if any) such as allergic reactions, gastrointestinal symptoms (e.g. bloating, constipation), and neurological effects (e.g. headache, drowsiness, euphoria)?
2. What is usability experience for patients using the Callavid drug-device combination compared to pessaries (i.e. Cyclogest 400 mg)?
3. How do serum progesterone levels vary within participants when using 400 mg progesterone delivered via the Callavid drug-device combination compared to Cyclogest 400 mg, and what are the implications of this variability for dose-response relationships and future trial design?

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Clinical diagnosis of luteal phase insufficiency on the basis of one of the following:
* Spotting before first day of heavy menstrual bleeding
* Short time between ovulation and menstruation
* Symptoms of progesterone insufficiency
* Aged 18 - 45 years
* Experienced at least one previous miscarriage

Exclusion Criteria:

* Positive pregnancy test
* Currently breastfeeding
* Allergies or contraindications to excipients / progesterone pessaries
* Current or history of previous condition where hormone treatments are contraindicated e.g. breast cancer
* Individuals who lack capacity to consent to the trial
* Individuals who have an inability to comply with the trial procedures (e.g. cannot attend hospital for trial visits)
* Inability to understand English

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Assigned female at birth.
Enrollment: 20 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Adverse events recorded from 400 mg progesterone Callavid | From treatment up to 24 hours after the last dose
  Any grade of adverse events, specifically allergy, gastrointestinal (bloating, constipation), neurological (headache, drowsiness, euphoria) according to Common Terminology Criteria for Adverse Events (CTCAE).

SECONDARY OUTCOMES:
PROMIS Anxiety questionnaire | Day 1 and day 7 of treatment in each round (3 rounds total)
  PROMIS short 4-item anxiety fear instrument
Acceptability questionnaires | Day 1 and day 7 of treatment in each round (3 rounds total)
  User acceptability questionnaires on 400mg progesterone Callavid
Semi-structured user experience interviews | day 7
  Semi-structured interviews with participants after completion of the crossover rounds.
Delivery of vaginal progesterone into the blood at 2 hour and 3 hour wear | Multiple time points on Day 1 and Day 7 of each treatment
  The serum progesterone levels at time 0, 3- and 6-hour after the first dose on day 1 and the thirteenth dose which is on day 7 each round of treatment are measured. Progesterone levels are measured for both 400 mg progesterone Callavid and 400 mg Cyclogest.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Coventry & Warwickshire NHS Trust, Coventry, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided